CLINICAL TRIAL: NCT01253551
Title: A Phase 1, Open-label, Randomized, Crossover Study in 20 Healthy Subjects to Investigate the Potential Pharmacokinetic Interaction Between Telaprevir and Raltegravir, Both at Steady-state
Brief Title: VX-950HEP1001 - Drug-drug Interaction Study Between Telaprevir and Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017608; VX-950HEP1001
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: VX-950HEP1001; hepatitis; telaprevir; raltegravir; crossover; healthy volunteers; VX-950.
MeSH Terms: conditions — Hepatitis C; Hepatitis

ARMS (2):
- 001 (Experimental): Treatment sequence AB Treatment A: telaprevir 750 mg every 8 hours on Days 1 to 6 with a morning dose on Day 7. Treatment B: raltegravir 400 mg twice a day on Days 1 to 10 and telaprevir 750 mg every 8 hours on Days 5 to 10 with a morning dose of raltegravir and a morning and afternoon dose of telaprevir on Day 11.
  Interventions: Drug: Treatment sequence AB
- 002 (Experimental): Treatment sequence BA Treatment A: telaprevir 750 mg every 8 hours on Days 1 to 6 with a morning dose on Day 7. Treatment B: raltegravir 400 mg twice a day on Days 1 to 10 and telaprevir 750 mg every 8 hours on Days 5 to 10 with a morning dose of raltegravir and a morning and afternoon dose of telaprevir on Day 11.
  Interventions: Drug: Treatment sequence BA

INTERVENTIONS:
Drug: Treatment sequence AB — Treatment A: telaprevir 750 mg every 8 hours on Days 1 to 6, with a morning dose on Day 7. Treatment B: raltegravir 400 mg twice a day on Days 1 to 10 and telaprevir 750 mg every 8 hours on Days 5 to 10, with a morning dose of raltegravir, and a morning and afternoon dose of telaprevir on Day 11.
  Arms: 001
Drug: Treatment sequence BA — Treatment A: telaprevir 750 mg every 8 hours on Days 1 to 6, with a morning dose on Day 7. Treatment B: raltegravir 400 mg twice a day on Days 1 to 10 and telaprevir 750 mg every 8 hours on Days 5 to 10, with a morning dose of raltegravir, and a morning and afternoon dose of telaprevir on Day 11.
  Arms: 002

SUMMARY:
The purpose of this study is to confirm the absence of a clinically relevant interaction between telaprevir and raltegravir at steady-state.Telaprevir is being investigated for the treatment of chronic hepatitis C virus infection, and raltegravir is used to treat HIV infection.

DETAILED DESCRIPTION:
This is an open-label, randomized (the order in which you receive the treatment sessions is determined by chance, like tossing a coin), crossover (participants will receive different interventions sequentially during the trial) study in healthy participants to investigate the effect of telaprevir 750 mg, every 8 hours, on the pharmacokinetics (how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body) of raltegravir 400 mg, twice a day, and vice versa. The study population will consist of 20 healthy participants. Each individual participant will receive two treatments: Treatment A (telaprevir 750 mg, every 8 hours, alone, on Days 1 to 6, with a morning dose on Day 7) and Treatment B (raltegravir 400 mg, twice a day, on Days 1 to 10 and telaprevir 750 mg, every 8 hours, on Days 5 to 10, with a morning dose of raltegravir, and a morning and afternoon dose of telaprevir on Day 11). Half of the participants will receive first Treatment A and then Treatment B; the other half will receive first Treatment B and then Treatment A. There will be a washout period of at least 14 days between the 2 sessions. The screening period will be maximum 21 days; the treatment duration will be approximately 4.5 weeks, and the follow-up period will be 30 to 31 days. All study medication will be taken with food. On Day 7 of Treatment A and Day 11 of Treatment B, 9 blood samples will be taken for determination of the levels of telaprevir in the blood. On Days 4 and 11 of Treatment B, 10 blood samples will be taken for determination of the levels of raltegravir in the blood. Predose pharmacokinetic samples will be collected on other days during the treatment sessions. Safety and tolerability will be evaluated throughout the trial by evaluating results of blood and urine analyses, vital signs, physical examinations, electrocardiograms (electrical recording of the heart), drug and alcohol screenings, and by assessing how the participant is feeling. In Treatment A, participants will receive 2 oral tablets of telaprevir 375 mg every 8 hours on Days 1 to 6, with a morning dose on Day 7. In Treatment B, participants will receive 1 oral tablet of 400 mg raltegravir twice a day on Days 1 to 10 and 2 oral tablets of 375 mg telaprevir every 8 hours on Days 5 to 10, with a morning dose of raltegravir, and a morning and afternoon dose of telaprevir on Day 11.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram and clinical laboratory tests at screening
* A Body Mass Index of 18.0 to 30.0 kg/m2, extremes included
* Women must be postmenopausal for at least 2 years, be surgically sterile and should not be breastfeeding
* Men must agree to use 2 highly effective methods of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of the study drug
* Be non-smoking for at least 3 months prior to selection.

Exclusion Criteria:

* Current use of prescription medication, regular treatment with over-the-counter medications (to be stopped no less than 7 days prior to first intake of study medication) or consumption of herbal medications or dietary supplements, vitamins, grapefruit or grapefruit juice, apple juice or orange juice within 14 days before first intake of study medication
* Consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 glass of beer, 1 glass of wine, 25 mL shot of 40% spirit), consumption of alcohol 72 hours before or after study medication intake, consumption of an average of more than five 240 mL servings of coffee or other caffeinated beverages, eg, tea, cola per day
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use
* Received an investigational drug or vaccine or used an investigational medical device within 3 months or 5 half lives (whichever is longer) before the planned start of treatment or having participated previously in a study with telaprevir.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Blood levels of telaprevir and raltegravir when given alone versus when given together | Day 7 of Treatment A
Blood levels of telaprevir and raltegravir when given alone versus when given together | Day 4 of Treatment B
Blood levels of telaprevir and raltegravir when given alone versus when given together | Day 11 of Treatment B

SECONDARY OUTCOMES:
Percentage of participants with a given adverse event as a measure of safety and tolerability | From screening to end of study
Clinical laboratory abnormalities as a measure of safety and tolerability | At screening and at 5-7 days and 30-32 days after last dose (Treatment A or B)
Clinical laboratory abnormalities as a measure of safety and tolerability | On Days 1 and 7 (Treatment A)
Clinical laboratory abnormalities as a measure of safety and tolerability | On Days 1, 4, and 11 (Treatment B)
Vital signs observed values and changes from baseline as a measure of safety and tolerability | At screening and at 5-7 days and 30-32 days after last dose (Treatment A or B)
Vital signs observed values and changes from baseline as a measure of safety and tolerability | On Days 1 and 7 (Treatment A)
Vital signs observed values and changes from baseline as a measure of safety and tolerability | On Days 1, 4, and 11 (Treatment B)
Physical examination findings and changes from baseline as a measure of safety and tolerability | At screening, on Day -1 of Treatments A and B, and at 5-7 days and 30-32 days after last dose (Treatment A or B)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA